CLINICAL TRIAL: NCT05620758
Title: Clinical Effectiveness of a Laser Therapy in Patients With Temporomandibular Disorders (A Randomized Clinical Trial)
Brief Title: Laser Therapy and Temporomandibular Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMD_Laser_2022
Record Dates: First submitted 2022-11-10; First posted 2022-11-17 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: TMD
MeSH Terms: interventions — Lasers, Solid-State; Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Nd YAG laser (Experimental)
  Interventions: Other: Nd YAG laser
- Diode laser 980 nm (Experimental)
  Interventions: Other: diode laser (980 nm)
- Diode laser 940 nm (Experimental)
  Interventions: Other: diode laser (940 nm)
- Diode laser 660 nm (Experimental)
  Interventions: Other: diode laser (660 nm)
- Diode laser 635 nm (Experimental)
  Interventions: Other: diode laser (635 nm)

INTERVENTIONS:
Other: Nd YAG laser — patients from those diagnosed with TMD will receive Nd YAG laser 1064 nm
  Arms: Nd YAG laser
Other: diode laser (980 nm) — patients from those diagnosed with TMD will receive a diode laser (980 nm)
  Arms: Diode laser 980 nm
Other: diode laser (940 nm) — patients from those diagnosed with TMD will receive a diode laser (940 nm)
  Arms: Diode laser 940 nm
Other: diode laser (660 nm) — patients from those diagnosed with TMD will receive a diode laser (660 nm)
  Arms: Diode laser 660 nm
Other: diode laser (635 nm) — patients from those diagnosed with TMD will receive a diode laser (635 nm)
  Arms: Diode laser 635 nm

SUMMARY:
TMD involves a set of multiple clinical manifestations where the pain is prevalent. Treatment ideally should be noninvasive and innocuous such as photobiomodulation

ELIGIBILITY:
Inclusion Criteria:

* Pain at TMJ area.
* Pain at masseter and temporalis muscles.
* Age ranges between 20 and 40 years old.
* Presence of full or nearly full complement of natural teeth

Exclusion Criteria:

* Patients who have radiographic evidence of degenerative conditions of TMJ.
* Patients under current dental or physical therapy that could affect TMD.
* History of recent trauma.
* The presence of systemic diseases (i.e. rheumatoid arthritis, osteoarthritis).
* Pregnant and lactating females

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain | Baseline and 1 month
  Visual analogue scale of pain (VAS),using a 0-10-point scale 0 score means no pain" and score 10 means "worst pain
Chaneg in pressure pain threshold | Baseline and 1 month
  The pressure pain threshold measurements for the trapezius, infraspinatus, and extensor carpi radialis muscles were performed at the center of the upper trapezius, at a position 2-3 fingers below the center of the spine of scapula, and at a position 3-4 fingers below the lateral epicondyle of the humerus, respectively. The pressure pain threshold of the extensor indicis proprius was measured by pressing toward the medial side of the radius from a position 3 fingers above the radial styloid process. The investigator placed the digital pressure algometer on a site to be inspected and pressed against the tester in a vertical direction while increasing the force at a constant rate of 1 kg/cm2. The investigator instructed the subjects to express pain either by saying "ouch" or raising their hands when only slight pain was felt. After all 8 muscles were investigated, the subjects were allowed to rest for 5 min. This procedure was repeated a total of 3 times.
Change in Oral-health Related Quality of life (OHRQoL) | Baseline and 1 month
  The OHIP-14 has 14 questions related to the evaluation of OHRQoL. The responses were recorded in a 5-point Likert scale ranging from never to very often (score is 0 to 4). Then, we calculated the total scores of all domains, and a higher score indicated poor OHRQoL. The highest possible total score of all the OHIP-14 domains is 56

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt